CLINICAL TRIAL: NCT04963530
Title: Wear Evaluation of Antagonist Enamel to Monolithic Zirconia, Lithium Disilicate and Metal-ceramic Restorations. Prospective Randomised Study
Brief Title: Enamel Wear Evaluation in Patients With Different Ceramic Restorations
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Valencia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 186205
Record Dates: First submitted 2021-06-01; First posted 2021-07-15 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Wear, Tooth; Dental Wear; Prosthetic; Outcome
Keywords: Enamel wear; Monolithic zirconia; Lithium Disilicate; Metal-ceramic; Single crowns
MeSH Terms: conditions — Tooth Wear | interventions — Therapeutics; Metal Ceramic Alloys

STUDY DESIGN:
Intervention Model Description: This prospective study will include a sample "n" of 75 patients. Patients will be treated with single-tooth restorations with partial or complete veneering on the tooth. Depending on the material used to fabricate the restoration, 4 different groups will be differentiated: monolithic zirconia (group 1), metal-ceramic (group 2), lithium disilicate (group 3) and natural tooth (control group).
  The sample will be randomised into one of the different groups using the online randomisation software www.alazarinfo.es. All patients will be pseudonymised, assigning each patient a number from 1 to 75 according to the chronology of incorporation into the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Wear of antagonist teeth to monolithic zirconia restorations (Experimental): Evaluate enamel wear antagonist to monolithic zirconia restorations monitoring the short and medium-term volume loss and assessing the factors that may influence this wear.
  Interventions: Procedure: Treatment with monolithic zirconia restorations
- Wear of antagonist teeth to lithium disilicate restorations (Experimental): Evaluate enamel wear antagonist to lithium disilicate restorations monitoring the short and medium-term volume loss and assessing the factors that may influence this wear.
  Interventions: Procedure: Treatment with lithium disilicate restorations
- Wear of antagonist teeth to metalceramic restorations (Experimental): Evaluate enamel wear antagonist to metal ceramic restorations monitoring the short and medium-term volume loss and assessing the factors that may influence this wear.
  Interventions: Procedure: Treatment with metal ceramic restorations
- Wear of natural enamel (Experimental): Evaluate physiological enamel wear (control group) monitoring the short short and medium-term volume loss and assessing the factors that may influence this wear.
  Interventions: Procedure: No intervention

INTERVENTIONS:
Procedure: Treatment with monolithic zirconia restorations — Treatment with monolithic zirconia restorations on teeth (single crowns). The sample (75 patients) will be divided into three groups according to the ceramic material used: monolithic zirconia, lithium disilicate and metal ceramic.
  Arms: Wear of antagonist teeth to monolithic zirconia restorations
Procedure: Treatment with lithium disilicate restorations — Treatment with lithium disilicate restorations on teeth (single crowns). The sample (75 patients) will be divided into three groups according to the ceramic material used: monolithic zirconia, lithium disilicate and metal ceramic.
  Arms: Wear of antagonist teeth to lithium disilicate restorations
Procedure: Treatment with metal ceramic restorations — Treatment with metal ceramic restorations on teeth (single crowns). The sample (75 patients) will be divided into three groups according to the ceramic material used: monolithic zirconia, lithium disilicate and metal ceramic.
  Arms: Wear of antagonist teeth to metalceramic restorations
Procedure: No intervention — No intervention.
  Arms: Wear of natural enamel

SUMMARY:
The aim of this study is to evaluate the wear produced in the short and medium term by monolithic zirconia, metal-ceramic and lithium disilicate restorations on the antagonist natural enamel in patients with fixed prostheses, assessing the factors that may influence this wear.

The investigators will also analyse whether the wear of the tooth antagonistic to the different restorations differs significantly with respect to the wear of the natural tooth (control group). The null hypothesis is that there are no significant differences.

DETAILED DESCRIPTION:
The study will be carried out on patients who will be candidates for treatment with full coverage restorations on teeth (single crowns). These crowns will be made of one of the following materials: monolithic zirconia, lithium disilicate or metal-ceramic, which will be cemented according to the guidelines defined in the scientific literature.

Inclusion criteria will be: patients in need of full coverage crowns on a first or second premolar or first or second molar in any arch, over 18 years of age, no contraindications for dental treatment, good oral hygiene, no periodontal disease or treated periodontal disease, absence of temporomandibular disorder and/or untreated habits or parafunctions.

The aim of this study is to evaluate the wear produced in the short and medium term by monolithic zirconia, metal-ceramic and lithium disilicate restorations on the antagonist tooth in patients with fixed prostheses, assessing the factors that may influence this wear.

The investigators will also analyse whether the wear of the tooth antagonistic to the different restorations differs significantly with respect to the wear of the natural tooth (control group). The null hypothesis is that there are no significant differences.

Once the treatment has been completed, the patient must attend routine check-ups in which a complete intraoral exploration, a scan and data collection for both arches will be carried out in order to analyse the following variables: wear of the antagonist tooth to ceramic restorations, wear of the restoration itself and physiological wear of the natural tooth. The same intervention will be carried out for the duration of the project, at the following time intervals: baseline (day of cementation of the restoration), 1 month, 6 months and annually. If an intraoral scanner is not available, silicone impressions will be made, which will be cast with plaster and scanned extraorally.

The investigators will work with a sample "n" of 75 patients, collected over the next two years. Depending on the material used to fabricate the restoration, 4 different groups will be differentiated: monolithic zirconia (group 1), metal-ceramic (group 2), lithium disilicate (group 3) and natural tooth (control group). The patients will be randomly distributed into the different groups using the online randomisation software www.alazarinfo.es.

ELIGIBILITY:
INCLUSION CRITERIA:

* Patients in need of single tooth restorations on posterior teeth.
* Age range: between 18 years of age.
* No contraindications for dental treatment.
* Good oral hygiene.
* No periodontal disease or treated periodontal disease.
* Absence of temporomandibular disorder and/or untreated habits or parafunctions.

Inclusion criteria for abutment teeth:

1. Posterior tooth requiring placement of a single tooth restoration. Restorability: with a crown:root ratio of at least 1:1.
2. The presence of an unrestored or minimally restored natural antagonist tooth (teeth with no more than a Class II restoration), in the same quadrant as the treated tooth (G1,2,3).
3. The presence of two unrestored or minimally restored antagonist teeth (in the same quadrants or on the contralateral side) (G4 or control).
4. Minimum height of the dental stump: 3mm.

EXCLUSION CRITERIA:

Exclusion criteria for abutment teeth:

1. Antagonist tooth with a full coverage restoration.
2. Opposing arch with fixed or removable partial denture.
3. Lack of occlusal contact points in the enamel of the control teeth.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Enamel volume loss | Through study completion, an average of two years
  Analyse volume loss of enamel antagonist to monolithic zirconia, lithium disilicate and metal ceramic restorations. The investigators will also analyse whether the wear of the tooth antagonistic to the different restorations differs significantly with respect to the physiological wear of the natural tooth (control group).

SECONDARY OUTCOMES:
Survival | Through study completion, an average of two years
  To compare the survival between monolithic zirconia, lithium disilicate and metal ceramic restorations.

CONTACTS AND LOCATIONS:
Overall Officials: Mª Fernanda Solá Ruiz, Dentistry, Principal Investigator — University of Valencia
Locations (1):
- Mª Fernanda Solá Ruiz, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-02-01): https://cdn.clinicaltrials.gov/large-docs/30/NCT04963530/Prot_SAP_000.pdf
  • Informed Consent Form (2021-02-01): https://cdn.clinicaltrials.gov/large-docs/30/NCT04963530/ICF_001.pdf